CLINICAL TRIAL: NCT04264650
Title: Long-term Effectiveness of an mHealth Intervention for Improving the Disease Knowledge and Physical Activity of Youth With Congenital Heart Disease: A Randomized Controlled Trial
Brief Title: Effectiveness of an mHealth Intervention for Youth With Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Chi-Wen Chen, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201603045RINA
Record Dates: First submitted 2020-02-09; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Congenital Heart Disease; Adolescent Behavior
MeSH Terms: conditions — Heart Defects, Congenital; Adolescent Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Standard care
- One active intervention group (Experimental): provided with COOL Passport, a mobile healthcare application
  Interventions: Behavioral: an mHealth intervention
- The other active intervention group (Experimental): provided with access to the Health Promotion Cloud system and use of game-based interactive platforms along with COOL Passport
  Interventions: Behavioral: an mHealth intervention

INTERVENTIONS:
Behavioral: an mHealth intervention — The Care & Organize Our Lifestyle (COOL) program, a self-regulation theory-based mHealth program
  Arms: One active intervention group; The other active intervention group

SUMMARY:
The aims of this study were to evaluate the long-term effectiveness of the Care & Organize Our Lifestyle (COOL) program, a self-regulation theory-based mHealth program, on improving disease knowledge and physical activity in youth with congenital heart disease (CHD). The COOL program is a 12-month randomized controlled trial that compared two active intervention groups to a standard-care control group (n = 47). Participants with simple and moderate CHD aged 15-24 years were recruited from pediatric or adult CHD outpatient departments. Participants in one active intervention group (n = 49) were provided with COOL Passport, a mobile healthcare application. Those in the other group (n = 47) were provided with access to the Health Promotion Cloud system and use of game-based interactive platforms along with COOL Passport. Outcomes were the Leuven Knowledge Questionnaire for CHD and the International Physical Activity Questionnaire-Taiwan Show-Card Version.

DETAILED DESCRIPTION:
Background: Mobile health initiatives may provide youth with congenital heart disease (CHD) relevant health information and a platform for managing the complex health care needs associated with undergoing transitional care.

Aims: To evaluate the long-term effectiveness of the Care & Organize Our Lifestyle (COOL) program, a self-regulation theory-based mHealth program, on improving disease knowledge and physical activity in youth with CHD.

Methods: The COOL program is a 12-month randomized controlled trial that compared two active intervention groups to a standard-care control group (n = 47). Participants with simple and moderate CHD aged 15-24 years were recruited from pediatric or adult CHD outpatient departments. Participants in one active intervention group (n = 49) were provided with COOL Passport, a mobile healthcare application. Those in the other group (n = 47) were provided with access to the Health Promotion Cloud system and use of game-based interactive platforms along with COOL Passport. Outcomes were the Leuven Knowledge Questionnaire for CHD and the International Physical Activity Questionnaire-Taiwan Show-Card Version.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with CHD by a pediatric cardiologist and qualifying as having simple or moderate CHD complexity according to the 2008 American College of Cardiology/American Heart Association guidelines;
* having a regular pulse;
* being 15-24 years of age;
* being conversant in Mandarin and Taiwanese;
* possessing a smartphone with Internet connection;
* agreeing to wear an exercise-monitoring wristband to record physiological data;
* agreeing to engage in exercises designed to test cardiopulmonary endurance;
* agreeing to participate in the study and sign an informed consent form for a relevant interview. For participants under 20 years of age, guardian approval by signing a written consent form was required.

Exclusion Criteria:

* having cognitive impairment to the extent of being noncommunicative;
* having CHD complicated with other congenital abnormalities;
* having undergone a cardiac catheter-related intervention or surgery within the past 6 months;
* being pregnant

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 143 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Cardiac disease knowledge | 12 months
  measured by the Leuven Knowledge Questionnaire for CHD

SECONDARY OUTCOMES:
Physical activity | 12 months
  measured by the International Physical Activity Questionnaire-Taiwan Show-Card Version

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Wen Chen, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin PJ, Fanjiang YY, Wang JK, Lu CW, Lin KC, Cheong IM, Pan KY, Chen CW. Long-term effectiveness of an mHealth-tailored physical activity intervention in youth with congenital heart disease: A randomized controlled trial. J Adv Nurs. 2021 Aug;77(8):3494-3506. doi: 10.1111/jan.14924. Epub 2021 Jun 21. PMID 34151444
- [Derived] Williams CA, Wadey C, Pieles G, Stuart G, Taylor RS, Long L. Physical activity interventions for people with congenital heart disease. Cochrane Database Syst Rev. 2020 Oct 28;10(10):CD013400. doi: 10.1002/14651858.CD013400.pub2. PMID 33112424